CLINICAL TRIAL: NCT01149980
Title: Randomized, 2-way Crossover, Bioequivalence Study of Citalopram Hydrobromide 40 mg Tablets and Celexa 40 mg Tablets Administered as 1 x 40 mg Tablet in Healthy Subjects Under Fed Conditions
Brief Title: Bioequivalence Study of Citalopram Hydrobromide Tablets 40 mg of Dr.Reddy's Laboratories Limited Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Dr.Ramakrishna Banagaru, Dr. Reddy's Laboratories Limited
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 30285
Record Dates: First submitted 2010-06-21; First posted 2010-06-24 (Estimated); Last update posted 2010-06-24 (Estimated); Status verified 2010-06

CONDITIONS: Healthy
Keywords: Bioequivalence; Crossover; Citalopram
MeSH Terms: interventions — Citalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Citalopram (Experimental): Citalopram Hydrobromide Tablets 40 mg of Dr.Reddy's
  Interventions: Drug: Citalopram Hydrobromide
- Celexa (Active Comparator): Celexa 40 mg Tablets of Forest Labs
  Interventions: Drug: Citalopram Hydrobromide

INTERVENTIONS:
Drug: Citalopram Hydrobromide — Citalopram Hydrobromide Tablets 40 mg of Dr.Reddy's Laboratories Limited
  Other Names: Celexa Tablets 40 mg

SUMMARY:
This is a bioequivalence study of Citalopram Hydrobromide Tablets 40 mg of Dr.Reddy's Laboratories Limited under fed conditions.

DETAILED DESCRIPTION:
randomized, 2-way crossover; bioequivalence study of citalopram hydrobromide 40 mg tablets and celexa 40 mg tablets administered as

1 x 40 mg tablet in healthy subjects under fed conditions.

ELIGIBILITY:
Inclusion Criteria:

Subjects enrolled in this study will be members of the community at large. The recruitment advertisements may use various media types (e.g. radio, newspaper, Anapharm Inc.Web site, Anaphann Inc. volunteers' data base). Subjects must meet all of the following criteria in order to be included in the study:

* Non-child-bearing potential female or simale, smokers and/or non-smoker, 18 years of age and older.
* Subjects capable of consent
* Non-child-bearing potential female subject:
* Post-menopausal state: absence of menses for 12 months prior to drug administration or hysterectomy with bilateral oophorectomy at least 6 months prior to drug administration.
* Surgically sterile: hysterectomy, bilateral oophorectomy, or tubal ligation at least 6 months prior to drug administration.

Exclusion Criteria:

* Subjects to whom any of the following applies will be excluded from the study:

  * Clinically significant illnesses within 4 weeks prior to the administration of the study medication.
  * Clinically significant surgery within 4 weeks prior to the administration of the study medication.
  * Any clinically significant abnormality found during medical screening.
  * Any reason which, in the opinion of the Medical Sub-Investigator, would prevent the subject from participating in the study.
  * Abnormal laboratory tests judged clinically significant.
  * Positive urine drug screen at screening.
  * Positive testing for hepatitis B, hepatitis C, or Human Immunodeficiency Virus HIV) at screening.
  * ECG abnormalities (clinically significant) or vital sign abnormalities (systolic blood pressure lower than 90 or over 140 mmHg, diastolic blood pressure lower than 50 or over 90 mmHg, or heart rate less than 50 or over 100 bpm)at screening.
  * Subjects with Body Mass Index (BMI) 2:30.0.
  * History of significant alcohol abuse within six months prior to the screening visit or any indication of the regular use of more than fourteen units of alcohol per week (1 Unit = 150 mL of wine, 360 mL of beer, or 45 mL of 40% alcohol).
  * History of drug abuse or use of illegal drugs: use of soft drugs (such as marijuana) within 3 months prior to the screening visit or hard drugs (such as cocaine, phencyclidine [PCP]and crack) within 1 year prior to the screening visit.
  * History of allergic reactions to citalopram hydrobromide or other related drugs.
  * History of allergic reactions to heparin.
  * Use of any drugs known to induce or inhibit hepatic drug metabolism (examples of inducers: barbiturates, carbamazepine, phenytoin, glucocorticoids, rifampin/rifabutin; examples of inhibitors: antidepressants, cimetidine, diltiazem, erythromycin, ketoconazole, Mono Amine Oxidase (MAO) inhibitors, neuroleptics, verapamil, quinidine) within 30 days prior to administration of the study medication.
  * Use of an investigational drug or participation in an investigational study within 30 days prior to administration of the study medication.
  * Clinically significant history or presence of any clinically significant gastrointestinal pathology (e.g. chronic diarrhea, inflammatory bowel diseases). Unresolved gastrointestinal symptoms (e.g. diarrhea, vomiting), liver or kidney disease, or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of the drug.
  * Any clinically significant history or presence of clinically significant neurological,endocrinal, cardiovascular, pulmonary, hematologic, immunologic psychiatric or metabolic disease.
  * Use of prescription medication (including hormone therapy) within 14 days prior to administration of study medication or over-the-counter products (including natural food supplements, vitamins, garlic as a supplement) within 7 days prior to administration of study medication, except for topical products without systemic absorption.
  * Smoking more than 25 cigarettes per day.
  * Any food allergy, intolerance, restriction or special diet that could, in the opinion of the Medical Sub-Investigator, contraindicate the subject's participation in this study.
  * A depot injection or an implant of any drug within 3 months prior to administration of study medication.
  * Donation of plasma (500 mL) within 7 days prior to drug administration. Donation or loss of whole blood prior to administration of the study medication as follows:
  * less than 300 mL of whole blood within 30 days,
  * 300 mL to 500 mL of whole blood within 45 days or
  * more than 500 mL of whole blood within 56 days prior to drug administration.
  * Consumption of food or beverages containing grapefruit (e.g. fresh, canned or frozen)within 7 days prior to administration of the study medication.
  * History of seizure disorder or bipolar affective disorder.
  * Active psychiatric diagnosis.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2003-10; Primary Completion 2003-11 (Actual); Study Completion 2003-11 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on Cmax and AUC parameters | 2 Months

CONTACTS AND LOCATIONS:
Overall Officials: Benoit Girard, M.D, Principal Investigator — Anapharm. Clinical Laboratory
Locations (1):
- Anapharm, Québec, Canada